CLINICAL TRIAL: NCT00092417
Title: Evaluation of the Safety and Tolerability of a Higher Potency Dose of Varicella Zoster Virus Vaccine Live (Oka/Merck)Among Adults 50 Years of Age or Older
Brief Title: Evaluation of the Safety and Tolerability of a Higher Potency Dose of an Investigational Vaccine Among Adults 50 Years of Age and Older (V211-009)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-009; 2004_075
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Results first posted 2010-06-10 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Higher Potency Dose
  Interventions: Biological: Comparator: Varicella Zoster Virus Vaccine
- 2 (Experimental): Lower Potency Dose
  Interventions: Biological: Comparator: Varicella Zoster Virus Vaccine

INTERVENTIONS:
Biological: Comparator: Varicella Zoster Virus Vaccine — Single 0.65 mL subcutaneous injection of higher potency zoster vaccine (~207,000 plaque-forming units [PFU]/0.65-mL dose)
  Arms: 1
Biological: Comparator: Varicella Zoster Virus Vaccine — Single 0.65 mL subcutaneous injection of lower potency zoster vaccine (~58,000 plaque-forming units [PFU]/0.65-mL dose)
  Arms: 2

SUMMARY:
This study compared the safety and tolerability profile of a higher potency investigational vaccine to that of the investigational vaccine at a lower potency dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals 50 years of age or older with a history of chickenpox who have not had herpes zoster

Exclusion Criteria :

* Preexisting conditions that might affect vaccine safety such as conditions that inhibit an immune response

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2003-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Tyring SK, Diaz-Mitoma F, Padget LG, Nunez M, Poland G, Cassidy WM, Bundick ND, Li J, Chan IS, Stek JE, Annunziato PW; Protocol 009 Study Group. Safety and tolerability of a high-potency zoster vaccine in adults >/= 50 or years of age. Vaccine. 2007 Feb 26;25(10):1877-83. doi: 10.1016/j.vaccine.2006.10.027. Epub 2006 Oct 30. PMID 17227688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 18 sites in the United States, Canada, and Europe
  Prime Therapy Period: 30-Oct-2003 to 07-Jun-2004
  Cutoff date for in-house data: 24-Aug-2004
Groups:
- Zoster Vaccine Higher Potency: Higher potency Zoster vaccine (approximately 207,000 plaque-forming units [PFU]), 1 subcutaneous 0.65 mL injection
- Zoster Vaccine Lower Potency: Lower potency Zoster vaccine (approximately 58,000 PFU), 1 subcutaneous 0.65 mL injection
Period: Overall Study
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Started | 464 (Started Period Group 1) | 234 (Started Period Group 2)
Vaccinated | 461 (3 participants were allocated,not vaccinated; they are not reported in the Baseline Characteristics) | 234
Completed | 459 (Received the higher potency zoster vaccine & completed 42 days of safety follow-up post vaccination) | 233 (Received the lower potency zoster vaccine & completed 42 days of safety follow-up post vaccination)
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency | Total
Number analyzed (Participants) | 461 | 234 | 695
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.16) | 65.6 (9.69) | 65.4 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 134 | 416
  Male | 179 | 100 | 279
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10 | 6 | 16
  Black | 6 | 4 | 10
  Hispanic American | 10 | 8 | 18
  Multi-Racial | 1 | 2 | 3
  Native American | 2 | 0 | 2
  White | 432 | 214 | 646

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaccine-related Serious Clinical Adverse Experiences (SAEs)
Description: The incidence of vaccine-related SAEs occurring Day 1 through Day 42 postvaccination. Whether a serious clinical adverse experience occurring Day 1 through Day 42 postvaccination was vaccine-related was determined by the investigator who was a qualified physician . The difference in the risk of developing a vaccine-related SAE between the two groups was compared at the 2-sided 0.05 level.
Time Frame: Day 1-42 post vaccination
Population: The population for the primary safety analysis consisted of all vaccinated participants who had safety follow-up data.
Measure: Number; unit: Participants
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Number analyzed (Participants) | 459 | 234
Participants
  With vaccine-related SAEs | 0 | 0
  Without vaccine-related SAEs | 459 | 234

2. Primary Outcome: Number of Participants With Moderate or Severe Injection-site Pain/Tenderness/Soreness or Swelling (> 2 Inches at Largest Diameter)
Time Frame: Day 1-5 postvaccination
Population: The population for the primary safety analysis consisted of all vaccinated participants who had safety follow-up data.
Measure: Number; unit: Participants
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Number analyzed (Participants) | 459 | 234
Participants
  With moderate or severe injection-site reaction | 79 | 21
  Without moderate or severe injection-site reaction | 380 | 213

3. Other Pre Specified Outcome: Number of Participants With Varicella or Varicella-like Noninjection-site Rashes, Nondermatomal in Distribution With >100 Lesions
Description: Noninjection-site rash Day 1 through Day 42 postvaccination was reported by the participant to the investigator and confirmed to be varicelliform rash by the study physician and polymerase chain reaction (PCR).
Time Frame: Day 1-42 postvaccination
Population: The population for the safety analyses consisted of all vaccinated participants who had safety follow-up data.
Measure: Number; unit: Participants
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Number analyzed (Participants) | 459 | 234
Participants
  With varicella or rash, varicelliform | 0 | 0
  Without varicella or rash, varicelliform | 459 | 234

4. Other Pre Specified Outcome: Number of Participants With Herpes Zoster (HZ) or HZ-like Rashes
Description: Noninjection-site rash Day 1 through Day 42 postvaccination was reported by the participant to the investigator and confirmed to be zosteriform rash by the study physician and polymerase chain reaction (PCR).
Time Frame: Day 1-42 postvaccination
Population: The population for the safety analyses consisted of all vaccinated participants who had safety follow-up data.
Measure: Number; unit: Participants
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Number analyzed (Participants) | 459 | 234
Participants
  With zoster or rash, zosteriform | 3 | 3
  Without zoster or rash, zosteriform | 456 | 231

5. Other Pre Specified Outcome: Number of Participants With Fevers ≥101.0°F [≥38.3°C]
Description: Maximum reported oral or equivalent temperature ≥101.0°F [≥38.3°C] was reported Day 1 through Day 21 postvaccination.
Time Frame: Day 1-21 postvaccination
Population: The population for the safety analyses consisted of all vaccinated participants who had safety follow-up data. 5 participants in the Zoster Vaccine Higher Potency group and 3 participants in the Zoster Vaccine Lower Potency group were not included in this analysis since these participants were without a follow-up.
Measure: Number; unit: Participants
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Number analyzed (Participants) | 456 | 231
Participants
  With max oral temp ≥101.0°F (≥38.3°C) | 4 | 2
  With max oral temp <101.0°F (<38.3°C) | 452 | 229

ADVERSE EVENTS:
Time Frame: Day 1 - 42 postvaccination
Description: Daily temperature readings, injection-site adverse experiences, rashes, and other adverse experiences were recorded by the participant on a Vaccination Report Card which was reviewed 42 days after vaccination.
  Number of participants at risk included randomized participants who had follow-up after at least one dose of vaccination.
Arm/Group | Zoster Vaccine Higher Potency | Zoster Vaccine Lower Potency
Serious Adverse Events (participants affected / at risk) | 4/459 | 1/234
Other Adverse Events (participants affected / at risk) | 296/459 | 141/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoster Vaccine Higher Potency (N=459) | Zoster Vaccine Lower Potency (N=234)
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoster Vaccine Higher Potency (N=459) | Zoster Vaccine Lower Potency (N=234)
Headache (Nervous system disorders) | 43 | 16
Injection Site Erythema (General disorders) | 227 | 111
Injection Site Pain (General disorders) | 217 | 91
Injection Site Pruritus (General disorders) | 58 | 21
Injection Site Swelling (General disorders) | 189 | 77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.